CLINICAL TRIAL: NCT05162092
Title: Effects of Vestibular Stimulation on Motor Function and Balance in Children With Hypotonic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 893
Record Dates: First submitted 2021-11-16; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hypotonic Cerebral Palsy
Keywords: vestibular stimulation; motor function; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: study participants will be randomized in two groups,conventional physiotherapy group and intervention group
Who Masked: Care Provider, Outcomes Assessor
Masking Description: double (care provider ,outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): training duration for each session is 30 mints with 5 mints rest and it includes passive soft tissue elogation of tight muscles,lower limb resistance exercises,movement transition,balance board standing ,walking and stair climbing
  Interventions: Other: Conventional physiotherapy
- Group B (Experimental): It included passive soft tissue elongation of tight muscles,lower limb resistance exercises,movement transition,balance board standing ,walking and stair climbing and Vestibular Stimulation exercises such as Swinging in standing in all directions, trampoline jumps, rocking movement in rocking chair, gaze stabilization exercises and visual pursuit exercises under supervision.
  Interventions: Other: Vestibular stimulation with conventional physiotherapy

INTERVENTIONS:
Other: Conventional physiotherapy — Participants will be given Conventional Physiotherapy. It included Passive Soft tissue elongation of tight muscles, Lower limb resistance exercises, Movement transitions, balance board and foam board standing, walking and stair climbing.
  Arms: Group A
Other: Vestibular stimulation with conventional physiotherapy — Participants in group B will be given conventional physiotherapy and vestibular stimulation exercises. It included conventional is same as given to the conventional and Vestibular Stimulation
  Arms: Group B

SUMMARY:
my study base on 2groups with total sample size 68 patients .group A conventional physiotherapy group in which the duration of session is 30 mints with 5 mints rest .include soft tissue elogation of tight muscles,lowerlimb resistance exercise,movement transitions balance board standing walking and stair climbing.for group b (conventional physiotherapy and vestibular stimulation exercises)30 mints with 10 mints rest.same physiotherpy exercise re given with vestibular stimulation exercises include swinging in standing in all diection,trampoline jump,rocking movement in rocking chair gaze stabilization exercises and visual pursuit exercises

DETAILED DESCRIPTION:
my study base on 2groups with total sample size 68 patients .group A conventional physiotherapy group in which the duration of session is 30 mints with 5 mints rest .include soft tissue elogation of tight muscles,lowerlimb resistance exercise,movement transitions balance board standing walking and stair climbing.for group b (conventional physiotherapy and vestibular stimulation exercises)30 mints with 10 mints rest.same physiotherpy exercise re given with vestibular stimulation exercises include swinging in standing in all diection,trampoline jump,rocking movement in rocking chair gaze stabilization exercises and visual pursuit exercises under supervisio. and use 2 scales,pediatric balance scale and gross motor scale re used for taking data .

ELIGIBILITY:
Inclusion Criteria:

* age range from 5-10 years.
* both male/female
* have good head control
* hypotonic cerebral palsy
* able to maintained ring sitting position

Exclusion Criteria:

* children will not respond to visual and auditory stimuli due to blindness or deafness or sever mental retardation
* children with un controlled convulsion or vp shunt
* children with severe medical problems children with orthopedic condition

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2021-07-04 (Actual); Primary Completion 2022-03-04 (Estimated); Study Completion 2022-03-04 (Estimated)

PRIMARY OUTCOMES:
Gross motor | 5 weeks
  A motor skill is a function, which involves precise movement of muscles with the intent to perform a specific act. Most purposeful movement requires the ability to "feel" or sense what one's muscles are doing as they perform the act. To measure the gross motor, gross motor function classification system is used. Gross motor function measure: The gross motor skill (sitting walking) of children and young people with cerebral palsy can be categorized into different level using a tool called gross motor function classification scale. Gross motor function scale has total of five levels. Level 1 is the lowest while level 5 is the highest. Higher level means worst outcome
Balance: | 5 weeks
  A biological system that enables us to know where our bodies are in the environment and to maintain a desired position. Normal balance depends on information from the inner ear, other senses (such as sight and touch) and muscle movement. To measure the balance, pediatric balance scale is used. Pediatric Balance Scale: The pediatric balance scale is modified version of Berg Balance that is used to assess functional balance skill in school-aged children they have 14 components and a total of 56 score. The minimum score is 0 and 56 is the maximum score. Higher score means good outcome

CONTACTS AND LOCATIONS:
Overall Officials: bilal umer, Principal Investigator — University of Lahore; anam naz, Principal Investigator — University of Lahore
Locations (1):
- Mahwash Zulfiqar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No